CLINICAL TRIAL: NCT00768456
Title: Lokal Infiltrations Analgesi Med Ropivakain 0,5 % Versus Placebo VED Vaginal Hysterektomi: ET Prospektivt Randomiseret, Dobbeltblind ET, Placebo-kontrolleret Studie
Brief Title: Local Infiltration Analgesia With Ropivacaine Versus Placebo in Vaginal Hysterectomy: a Randomized, Double-Blind Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Billy B Kristensen, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: H-C-2008-030
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2008-07

CONDITIONS: Pain, Postoperative; Postoperative Nausea and Vomiting
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Local infiltration with Ropivacaine
  Interventions: Drug: Ropivacaine 0.5 %
- 2 (Placebo Comparator): Local infiltration with Placebo (NaCl)
  Interventions: Drug: Isotonic NaCl

INTERVENTIONS:
Drug: Ropivacaine 0.5 % — Local Infiltration with Ropivacaine 0.5 %
  Arms: 1
Drug: Isotonic NaCl — Local Infiltration with NaCl
  Arms: 2

SUMMARY:
The purpose of this study is to compare systematic local infiltration with Ropivacaine 0.5 % vs. Placebo in patients undergoing vaginal hysterectomy.

The hypothesis is that systematic local infiltration will reduce postoperative pain and postoperative opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* eligible for elective vaginal hysterectomy
* able to speak and understand Danish
* able to give informed consent

Exclusion Criteria:

* alcohol or medical abuse
* allergies to local anesthetics
* age < 18 yrs.
* intolerance to opioids

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 32 h

SECONDARY OUTCOMES:
PONV | 32 h

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark